CLINICAL TRIAL: NCT06135688
Title: Effects of Lidocaine Bolus and Continuous Infusion on Bispectral Index Values and Spectrum During Maintenance of Total Intravenous Anesthesia With Target Controlled Infusion (Schnider Model)
Brief Title: Effects of Lidocaine Bolus and Infusion on Bispectral Index Values and Spectrum During Anesthesia Maintenance
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Federico Linassi, MD, principal investigator, University of Padova
Other Study IDs: LidoMAST
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia Brain Monitoring; Lidocaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lidocaine has been shown to increase the hypnotic effects of Propofol, however no trials shows the effects on Bispectral Index Values (BIS) and spectral analysis during total intravenous anesthesia maintenance delivered with target controlled infusion (TCI) with stable Concnetration at the effector site of Propofol (CeP)

DETAILED DESCRIPTION:
Lidocaine has been shown to increase the hypnotic effects of Propofol, however no trials shows the effects on Bispectral Index Values (BIS) and spectral analysis during total intravenous anesthesia maintenence delivered with target controlled infusion (TCI) with stable concentration at the effector site of Propofol (CeP).

Aim of this study is to analyze BIS values and power spectrum before and after a lidocaine bolus (1,5 mg/kg delivered in 10 minutes) and a subsequent continuous infusion (1,5 mg/kg/min for 30 minutes) delivered at anesthetist's discretion for postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Undergo general anesthesia with Target Controlled Infusion of Propofol (Schnider model) and Remifentanil (Minto model) and Lidocaine bolus and continuous infusion for a total of 40 minutes.

Exclusion Criteria:

* Neurological disease
* Psychiatric disease
* Obesity

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women undergoing brast cancer surgery with general anesthesia with Propofol and Remifentanil TCI, and Lidocaine bolus and infusion for postoperative pain will be included.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-11-18 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Correlation between BIS values and power spectrum before and after lidocaine administration | We collect data about propofol concentration (ng/ml)and BIS values during general anaesthesia. We will collect BIS and TCI Propofol values during all the duration of anesthesia, form the start o anesthesia until the emergence from anesthesia
  Patients will receive during anesthesia maintenance a lidocaine bolus of 1,5 mg/kg delivered in 10 minutes and a lidocaine continuous infusion of 1,5 mg/kg/h for 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Treviso Regional Hospital, Treviso, TV, Italy